CLINICAL TRIAL: NCT06293885
Title: PLeurodesis Using Hypertonic Glucose Administration to Treat Post-operative Air Leaks Following Lung Resection Surgery (PLUG): Phase II Randomized Feasibility Trial
Brief Title: Pleurodesis Using Hypertonic Glucose
Acronym: PLUG-II
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Mehdi Qiabi, Thoracic Surgeon, Assistant Professor, Western university, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLUG-II
Record Dates: First submitted 2024-02-25; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Air Leak From Lung
Keywords: air leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D50 (Experimental): A solution of 50% glucose will be injected into the pleural space on the first and possibly the second day after surgery. The injection will be administered through the chest tube, which is already in place.
  Interventions: Drug: Dextrose 50
- Standard of care (Active Comparator): monitor air leak, if the air leak continues on post-operative day #5, a talc pleurodesis may be given.
  Interventions: Other: Standard of Care - No Dextrose 50

INTERVENTIONS:
Drug: Dextrose 50 — a solution of 50% glucose (D50) will be injected into your pleural space
  Other Names: D50
  Arms: D50
Other: Standard of Care - No Dextrose 50 — Standard of Care
  Arms: Standard of care

SUMMARY:
Air leaks from unhealed lung tissue following lung resection for benign or malignant lesions are one of the most common complications following thoracic surgery, occurring after 10% of major lung resections. The purpose of this study is to investigate the efficacy of intrapleural administration of Dextrose 50% to resolve air leaks after pulmonary resection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing scheduled pulmonary lobar or sublobar resection for cancer
* Presence of air leak on postoperative day 1 of at least 100 mL/min, as documented on the digital drainage system

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Prolonged Air Leak | 5 days postoperatively
  Prolonged Air Leak

SECONDARY OUTCOMES:
Duration of Chest Tubes | immediately after the surgery
  Duration of Chest Tubes
Home with Chest Tube | immediately after the surgery
  Home with Chest Tube (y/n)

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada